CLINICAL TRIAL: NCT02061124
Title: Effect of Bile Acid Sequestration on Postprandial GLP-1 Secretion, Glucose Homeostasis and Gut Microbiota
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Gentofte, Copenhagen (Other)
Collaborators: Sanofi (Industry)
Responsible Party: Principal Investigator, Andreas Brønden, MD, University Hospital, Gentofte, Copenhagen
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: H-2-2013-148
Record Dates: First submitted 2014-02-06; First posted 2014-02-12 (Estimated); Last update posted 2015-11-23 (Estimated); Status verified 2015-11

CONDITIONS: Type 2 Diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Sevelamer

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (4):
- T2DM, sevelamer (Active Comparator): Patients with type 2 diabetes treated with sevelamer
  Interventions: Drug: Sevelamer 1600 mg TID for 7 days
- T2DM, placebo (Placebo Comparator): Patients with type 2 diabetes treated with placebo
  Interventions: Drug: Placebo 1600 mg TID for 7 days
- Healthy subjects, sevelamer (Active Comparator): Healthy subjects treated with sevelamer
  Interventions: Drug: Sevelamer 1600 mg TID for 7 days
- Healthy subjects, placebo (Placebo Comparator): Healthy subjects treated with placebo
  Interventions: Drug: Placebo 1600 mg TID for 7 days

INTERVENTIONS:
Drug: Sevelamer 1600 mg TID for 7 days
  Arms: Healthy subjects, sevelamer; T2DM, sevelamer
Drug: Placebo 1600 mg TID for 7 days
  Arms: Healthy subjects, placebo; T2DM, placebo

SUMMARY:
Accumulating evidence suggests that bile acids and bacteria in our intestines may constitute essential components in the complex mechanisms regulating gut hormone secretion and glucose homeostasis. At the same time, bile acids and gut bacteria are interdependent. Thus, it is likely that modification of the enterohepatic circulation of bile acids can lead to changes in gut hormone secretion or gut bacteria composition and consequently affect glucose homeostasis.

The current study is a human interventional study with 7-day ingestion of a bile acid sequestrant or placebo, preceded and followed by meal tests and faecal sampling. The aim is to examine how (and if) bile acid sequestration can influence postprandial glucagon-like peptide-1 (GLP-1) secretion, gut microbiota and glucose homeostasis in patients with type 2 diabetes and healthy individuals. As a tool to sequester bile acids we will use sevelamer, a phosphate binding resin used in the treatment of hyperphosphataemia in adult patients with chronic kidney disease. Surprisingly, sevelamer was recently shown to improve glycaemic control in patients with chronic kidney disease and type 2 diabetes.

The investigators hypothesize that higher luminal concentrations of bile acids in the distal gut will elicit changes in the postprandial gut hormone secretion and gut bacteria composition. The current study will help to clarify this hypothesis and improve our general understanding of the association between bile acid circulation and signalling, gut hormone secretion, gut bacteria and glucose metabolism.

ELIGIBILITY:
Inclusion Criteria:

Both groups

* Caucasian ethnicity
* Normal haemoglobin
* Age above 35 years and below 80 years
* Informed and written consent
* BMI > 23 kg/m2 and <35 kg/m2

Patients with type 2 diabetes

* Type 2 diabetes for at least 3 months
* Diagnosed according to the criteria of the World Health Organization (WHO)

Healthy Subjects

* Normal fasting plasma glucose (FPG) <6.5 mM and
* Normal glycated haemoglobin (HbA1c) <6.0 %

Exclusion Criteria:

Both groups

* Liver disease (alanine aminotransferase (ALAT) and/or serum aspartate aminotransferase (ASAT) >2 times normal values) or history of hepatobiliary disorder
* Gastrointestinal disease, previous intestinal resection, cholecystectomy or any major intra-abdominal surgery
* Hypo- or hyperphosphataemia
* Nephropathy (serum creatinine >150 µM and/or albuminuria
* Treatment with medicine that cannot be paused for 12 hours
* Intake of antibiotics six months prior to study
* Hypo- or hypercalcaemia
* Hypo- and hyperthyroidism
* Treatment with oral anticoagulants
* Active or recent malignant disease
* Any treatment or condition requiring acute or sub-acute medical or surgical intervention
* Lack of effective birth control in premenopausal women
* Positive pregnancy test on study days in premenopausal women
* Tobacco smoking
* Any condition considered incompatible with participation by the investigators

Patients with type 2 diabetes

* Treatment with insulin
* Treatment with incretin-based therapy

Healthy Subjects

* Diabetes or
* prediabetes (fasting plasma glucose levels >6.5 mM or HbA1c >6.0%)
* First-degree relatives with diabetes

Ages: 35 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2014-02; Primary Completion 2015-10 (Actual); Study Completion 2015-10 (Actual)

PRIMARY OUTCOMES:
Incremental and total area under the Concentration-Time Curve (AUC 0-240 min) | -30, -15, 0, 10, 20, 30, 45, 60, 90, 120, 180, 240 min on study days 1 and 7 (meal tests start at 0 min)
  Postprandial responses of glucagon-like peptide-1 (GLP-1)

SECONDARY OUTCOMES:
Incremental and total area under the Concentration-Time Curve (AUC 0-240 min) | -30, -15, 0, 10, 20, 30, 45, 60, 90, 120, 180, 240 min on study days 1 and 7 (meal tests start at 0 min)
  Postprandial responses of various other gut hormones

OTHER OUTCOMES:
Blood analysis | Fasting status on study days 1 and 7
  Lipids
Blood analysis | Fasting status on study days 1 and 7
  Inflammatory and metabolic markers
Faecal samples | Prior to study days 1 and 7
  Gut microbiota composition
Blood analysis of paracetamol | -30 min to 240 min (ingestion of meal at 0 min) on study days 1 and 7
  Assessment of gastric emptying
Bodyweight | Fasting state on study days 1 and 7
Indirect calorimetry | -30 min to 240 min (ingestion of meal at 0 min) on study days 1 and 7
  Basal metabolic rate
Ultrasound measurements | -30 min to 240 min (ingestion of meal at 0 min) on study days 1 and 7
  Gall bladder volume
Visual analog scale score | -30 min to 240 min (ingestion of meal at 0 min) on study days 1 and 7
  Appetite

CONTACTS AND LOCATIONS:
Locations (1):
- Diabetes Research Division, Gentofte Hospital, Copenhagen, Hellerup, Denmark